CLINICAL TRIAL: NCT03185143
Title: Randomized, Double-Blind, and Placebo-Controlled Study to Assess a Single Dose of Low-Dose Naltrexone and Acetaminophen Combination Versus Sumatriptan in the Acute Treatment of Migraine With Nausea
Brief Title: Low-Dose Naltrexone and Acetaminophen Combination and Sumatriptan in the Acute Treatment of Migraine With Nausea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Allodynic Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANODYNE-2
Record Dates: First submitted 2017-06-08; First posted 2017-06-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2018-05

CONDITIONS: Migraine With and Without Aura
MeSH Terms: interventions — Naltrexone; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Naltrexone and Acetaminophen Combination (Experimental)
  Interventions: Drug: Naltrexone and Acetaminophen Combination
- Sumatriptan 100 mg (Active Comparator)
  Interventions: Drug: Sumatriptan 100 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone and Acetaminophen Combination — Treat a single Qualified Migraine attack.
  Arms: Naltrexone and Acetaminophen Combination
Drug: Sumatriptan 100 mg — One capsule contains Sumatriptan 100 mg and one capsule contains a sham for component B taken together to treat a single Qualified Migraine attack.
  Arms: Sumatriptan 100 mg
Drug: Placebo — One capsule contains a sham for component A and one capsule contains a sham for component B taken together to treat a single Qualified Migraine attack.
  Arms: Placebo

SUMMARY:
This proof-of-concept study compares side-by-side low-dose naltrexone and acetaminophen combination to sumatriptan in the acute treatment of migraine.

DETAILED DESCRIPTION:
The study consists of a screening visit, outpatient treatment of a moderate or severe migraine attack with a single dose of the study drug within 8 weeks, and End-of-Study Visit 2-7 days after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 65 years of age.
2. History of migraine with or without aura according to the International Classification of Headache Disorders (ICHD)-3rd edition (beta version) for at least one-year with first migraine prior to age 50.
3. Migraine-associated nausea with ≥half the migraine attacks.
4. 2 - 8 migraines per month in each of the previous 3 months.
5. The patient is able to complete study questionnaires, comply with the study requirements and restrictions, and willing to provide written informed consent and authorize HIPAA.
6. The female patient who is premenopausal or postmenopausal less than 1 year, or have not had surgical sterilization (i.e., tubal ligation, partial or complete hysterectomy) must have a negative urine pregnancy test, be non-lactating, and commit to using 2 methods of adequate and reliable contraception throughout the study and for 28 days after taking the last dose of the study drug (e.g., barrier with additional spermicidal, intra-uterine device, hormonal contraception). Male patients must be surgically sterile or commit to the use of 2 different methods of birth control during the study and for 28 days after the study.ice, hormonal contraception).

Exclusion Criteria:

1. The patient in the opinion of the investigator may have medication-overuse headaches (as defined by ICHD - 3 beta criteria for medication-overuse headache) during the preceding 3 months.
2. The patient in the opinion of the investigator has chronic migraine (as defined by ICHD - 3 beta criteria for chronic migraine) during the preceding 3 months.
3. History of cluster headaches or neurologically complicated migraine (hemiplegic, basilar, retinal, ophthalmoplegic).
4. Initiation or change in medications with possible migraine prophylactic effects during 3 months before inclusion into the trial (E.g., calcium channel blockers, tricyclic antidepressants, beta-blockers, or Botox).
5. Use of opiates or barbiturates more than 3 days per month.
6. Any concurrent medical or psychiatric condition, this includes, but is not limited to chronic unstable debilitating diseases, significant renal or hepatic impairment.
7. The patient has a history within the previous 3 years of abuse of any drug, prescription, illicit, or alcohol.
8. The Female patient is pregnant or breast-feeding. The Male patient is not practicing 2 different methods of birth control with their partner during the study, and for 28 days after the investigational drug last dose or will not remain abstinent during the study, and for 28 days after the last dose.
9. The patient has known-hypersensitivity reaction to any of the components of the investigational drug.
10. Consumption of analgesic medication or muscle relaxants (including all benzodiazepines) for other conditions on a regular basis.
11. The patient has used emergency care treatment more than 3 times in the previous 6 months.
12. The patient has participated in another study with an investigational drug within 30 days prior to randomization and/or plan to participate during the study.
13. The patient has a history of congenital heart disease, cardiac arrhythmias, or cardiovascular disease, e.g., ischemic heart disease (e.g., stable angina pectoris, unstable angina, vasospastic angina, myocardial infarction or silent myocardial ischemia), cerebrovascular syndromes (e.g., strokes of any type or transient ischemic attacks), peripheral vascular disease, ischemic bowel disease, or Raynaud syndrome.
14. Uncontrolled hypertension (sitting >160 mmHg systolic pressure or >95mmHg diastolic pressure).
15. The patient, in the investigator's opinion, is likely to have unrecognized cardiovascular or cerebrovascular disease.
16. History of epilepsy. Allergy to sulfonamides.
17. Consumption of monoamine oxidase inhibitor (MAOI) drug, tricyclic antidepressant, selective serotonin reuptake inhibitor (SSRI) or Serotonin Noradrenaline Reuptake Inhibitor (SNRI).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
The proportion of patients having no headache pain at 2 hours. | 2 hours
  Measured by asking the patients to self-report the current status of their headache pain on a four-point Likert scale (i.e., 0=none, 1=mild, 2=moderate, 3=severe).
The proportion of patients having the absence of the most bothersome migraine-associated symptom at 2 hours. | 2 hours
  The most bothersome migraine-associated symptom is prospectively identified at baseline. It is measured by asking the patients to self-report the current status of their associated symptom as present or absent.

SECONDARY OUTCOMES:
The proportion of patients having the absence of nausea, photophobia, phonophobia, and neck/shoulder pain at 2 hours. | 24 and 48 hours
  Measured by asking the patients to self-report the current status of their associated symptoms as present or absent.
The proportion of patients who used rescue medications within 24 hours. | 24 hours
The proportion of patients who are "sustained pain-free" at 24-hours and 48-hours. | 48 hours.
  Defined as having no headache pain at 2 hours after the dose, with no use of rescue medication and no relapse of headache pain within 24 hours (24-hour sustained pain-free) or 48 hours (48-hour sustained pain-free) after administration of the investigational drug.
The proportion of patients who had headache pain relapse within 48 hours | 48 hours
  Defined as the return of headache of any severity within 48 hours after administration of the investigational drug, when the patient was pain-free at 2 hours after the administration of the investigational drug.
The proportion of patients who experienced adverse events | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Annette C. Toledano, M.D., Principal Investigator — Allodynic Therapeutics, Inc
Locations (1):
- Annette C. Toledano, M.D., North Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided